CLINICAL TRIAL: NCT05776199
Title: Sonoelastography, Tensiomyography and Mechanosensitivity Between Latent, Active and Control Trigger Points in Myofascial Trigger Points of the Levator Scapulae Muscle.
Brief Title: Myofascial Trigger Points of the Levator Scapulae Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, PhD., Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 03/23
Record Dates: First submitted 2023-03-06; First posted 2023-03-20 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Myofascial Pain Syndrome
Keywords: physiotherapies techniques; sonoelastography;; muscle tension; neck pain
MeSH Terms: conditions — Myofascial Pain Syndromes; Neck Pain | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic Compression group (Experimental): IC group with conservative technique in trigger points in levator scapulae muscle
  Interventions: Diagnostic Test: Sonoelastography, tensiomyography and mechanosensitivity
- Dry needling group (Active Comparator): Dry needling group with invasive technique in trigger points in levator scapulae muscle
  Interventions: Diagnostic Test: Sonoelastography, tensiomyography and mechanosensitivity

INTERVENTIONS:
Diagnostic Test: Sonoelastography, tensiomyography and mechanosensitivity — To observe the differences between the different trigger points of the levator scapulae muscle by means of different diagnostic options.

SUMMARY:
Chronic neck pain (CNP) is considered one of the most common musculoskeletal disorders worldwide and myofascial pain syndrome (MPS) is the most prevalent musculoskeletal disorder in the majority of the population. However, normal tissue contractility changes and the different types of myofascial trigger points (MTrPs) measured by tensiomography have not yet been studied. For this reason, the aim of our study is to determine the differences in pressure pain threshold (PPT), tensiomyography and sonoelastography between the palpation zone of control points with respect to active and latent MTrPs in the levator scapulae muscles of subjects with CNP. A single-blind descriptive cross-sectional study is conducted with a convenience sample of 60 points (20 active, 20 latent and 20 control points) on both sides of the subject in the levator scapulae muscles of individuals diagnosed with CNP.

The order of outcome measurements for each point was PPT, manual tension index sonoelastography and tensiomyography separated by 15 minutes. Objective contractile parameters were: contraction time (Tc), mean relaxation time (Tr), maximum radial displacement (Dm), holding time (Ts) and delay time (Td).

ELIGIBILITY:
Inclusion Criteria:

* Bilateral presence of at least one active trigger point.
* One control point and one latent trigger point in the levator scapulae muscles.
* Subjects aged between 18 and 65 years.
* Subjects diagnosed with chronic neck pain for more than 6 weeks.
* Signed informed consent to be able to participate in the study.

Exclusion Criteria:

* Previous treatment for chronic neck pain (within one year) or medical history with a diagnosis of neuropathy.
* Rheumatoid arthritis.
* Myopathy.
* Cognitive impairment or mental disability.
* Skin disorders.
* Pregnancy.
* Activity level of a high-level athlete.
* Medical conditions (fractures, structural deformities and neoplasms).
* Surgical interventions in the cervical-dorsal region or upper extremities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
manual tension index sonoelastography | 1 week
  Measurement of manual ultrasound transducer tension on the trigger point of the levator scapulae

SECONDARY OUTCOMES:
tensiomyography | 1 week
  Ultrasound transducer tensiomyography measurement of the levator scapulae trigger point
minimum intensity of a stimulus that elicits the sensation of pain (pressure pain threshold). | 1 week
  patient-tolerable pain at the trigger point of the levator scapulae muscle measured by algometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Myburgh C, Lauridsen HH, Larsen AH, Hartvigsen J. Standardized manual palpation of myofascial trigger points in relation to neck/shoulder pain; the influence of clinical experience on inter-examiner reproducibility. Man Ther. 2011 Apr;16(2):136-40. doi: 10.1016/j.math.2010.08.002. Epub 2010 Sep 1. PMID 20813576
- [Result] Tous-Fajardo J, Moras G, Rodriguez-Jimenez S, Usach R, Doutres DM, Maffiuletti NA. Inter-rater reliability of muscle contractile property measurements using non-invasive tensiomyography. J Electromyogr Kinesiol. 2010 Aug;20(4):761-6. doi: 10.1016/j.jelekin.2010.02.008. Epub 2010 Mar 16. PMID 20236839
- [Result] Sigrist RMS, Liau J, Kaffas AE, Chammas MC, Willmann JK. Ultrasound Elastography: Review of Techniques and Clinical Applications. Theranostics. 2017 Mar 7;7(5):1303-1329. doi: 10.7150/thno.18650. eCollection 2017. PMID 28435467
- [Result] Thomas K, Shankar H. Targeting myofascial taut bands by ultrasound. Curr Pain Headache Rep. 2013 Jul;17(7):349. doi: 10.1007/s11916-013-0349-4. PMID 23793988
- [Result] Park G, Kim CW, Park SB, Kim MJ, Jang SH. Reliability and usefulness of the pressure pain threshold measurement in patients with myofascial pain. Ann Rehabil Med. 2011 Jun;35(3):412-7. doi: 10.5535/arm.2011.35.3.412. Epub 2011 Jun 30. PMID 22506152
- [Result] Turo D, Otto P, Shah JP, Heimur J, Gebreab T, Zaazhoa M, Armstrong K, Gerber LH, Sikdar S. Ultrasonic characterization of the upper trapezius muscle in patients with chronic neck pain. Ultrason Imaging. 2013 Apr;35(2):173-87. doi: 10.1177/0161734612472408. PMID 23493615
- [Result] Koo TK, Guo JY, Brown CM. Test-retest reliability, repeatability, and sensitivity of an automated deformation-controlled indentation on pressure pain threshold measurement. J Manipulative Physiol Ther. 2013 Feb;36(2):84-90. doi: 10.1016/j.jmpt.2013.01.001. PMID 23499143